CLINICAL TRIAL: NCT03928041
Title: A Prospective, Non-comparative, Multi-center, Post-market Clinical Study to Evaluate the Safety and Performance of PEEK-OPTIMA™ HA Enhanced Interbody Cages for the Treatment of Degenerative Disc Disease and Spondylolisthesis in the Lumbar Spine
Brief Title: A Clinical Study to Evaluate Safety and Performance of PEEK-OPTIMA™ HA Enhanced Interbody Cages in the Lumbar Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Invibio Ltd (Industry)
Collaborators: Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CES01
Record Dates: First submitted 2019-04-16; First posted 2019-04-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Degenerative Disc Disease Lumbar; Spondylolisthesis, Grade 1
Keywords: Lumbar Degenerative Disc Disease; Spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis; Lymphoma, Follicular; Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: All subjects will be recruited and receive the EVOS-HA prospectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- single prospective study (Other): All subjects who are entered into this trial will receive the EVOS Lumbar Interbody System (EVOS- HA).
  Interventions: Device: Device: EVOS Lumbar Interbody System (EVOS-HA)

INTERVENTIONS:
Device: Device: EVOS Lumbar Interbody System (EVOS-HA) — All subjects will receive the EVOS Lumbar Interbody System (EVOS-HA) device if according to the investigators opinion they are clinically indicated to have surgery treatment for degenerative disc disease and spondylolisthesis.

SUMMARY:
The purpose of this trial is to collect clinical outcomes including radiographic and CT outcomes in patients who undergo interbody spinal fusion using the EVOS Lumbar Interbody System.

DETAILED DESCRIPTION:
This prospective, non-comparative, multi-center, post-market trial will evaluate the safety and efficacy of the PEEK-OPTIMA™ HA Enhance Interbody Cages System - EVOS- HA in patients suffering from degenerative disc disease and spondylolisthesis in the lumbar spine. The trial will capture clinical outcomes, radiographic and CT outcomes over a 24 month period post operatively. Two centers will be involved in the recruitment of 30 patients. All patients will be drawn from clinics which focus on this type of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Is the subject aged 18 years of age or older and skeletally mature?
* Does the subject have a primary diagnosis of symptomatic degenerative disc disease (DDD) or symptomatic degenerative disc disease (DDD) with spondylolisthesis (Grade 1) at one or two contiguous levels from L2 to S1?
* Does the subject have discogenic back pain with degeneration of the disc confirmed by medical history, radiographic examination and MRI (MRI must be obtained within the 6 months prior to subject surgery and radiographs obtained within 3 months prior to subject surgery)?
* Is the subject judged by the Investigator to be suitable for transforaminal lumbar interbody fusion (TLIF) surgery based on their medical history?
* Is the subject indicated for surgical treatment with the EVOS Lumbar Interbody System with autologous bone graft?
* Has the subject completed at least 6 months of conservative non-operative treatment without obtaining adequate symptomatic relief?
* If the subject is female and of childbearing age, do they have a negative pregnancy test (by Beta HCG qualitative analysis), or do they have a history of a surgical sterilisation, or a history of no menses in the past twelve months?
* Is the subject, in the opinion of the Investigator, able to understand this clinical study, co-operate with the procedures and are they willing to return to the hospital for all the required post-operative follow-ups?
* Is the subject able to give voluntary, written informed consent to participate in this clinical study and from whom consent has been obtained?

Exclusion Criteria:

* Has the subject undergone previous spinal surgery at the affected disc level(s), excluding discectomy and laminectomy procedures?
* Does the subject have evidence of tumour and/or malignant disease with resultant life expectancy of less than two years?
* Does the subject have known osteoporosis or severe osteopenia as determined by the Investigator?
* Does the subject have rheumatoid arthritis, ankylosing spondylitis or are they immunocompromised?
* Does the subject have a known allergy to the material used in the instrumentation?
* Does the subject have evidence of an active infection and/or do they have any condition that would compromise their participation and follow-up in this clinical study?
* Is the subject receiving any drug treatment that may affect bone metabolism?
* If the subject is female, are they pregnant or lactating?
* Is the subject a current smoker, or have they stopped smoking less than 6 months ago?
* Is the subject a known drug or alcohol abuser or do they have a baseline opioid use greater than 30 mg of morphine equivalent/day or do they have psychological disorders that could affect follow-up care or treatment outcomes?
* Is the subject currently enrolled in a clinical study?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Interbody fusion rate | 6 months post - operatively
  Interbody fusion will be graded in accordance with Cook et al. 2004 where bridging bone is graded along the superior and inferior interfaces separately in 25% increments.

SECONDARY OUTCOMES:
To measure how much pain the subject is in according to a pain scale - 0-10 | 6 weeks, 3, 6, 12 and 24 months post operatively
  Visual Analogue Scale for back and leg - 0 - 10 cm (no pain - worst possible pain)
To measure the Quality of Life of the subject according to a set list of questions: Questionnaire SF-12 | pre-operatively, 6 weeks, 3, 6, 12 and 24 months post operatively
  Questionnaire SF-12 collection of questions health related to assess vitality, physical functioning, bodily pain, general health perceptions, emotional and physical functioning, social and mental health. Patients will pick from a set list of answers for each health related question. The responses on each item are scored and summarized into Physical and Mental Health Composite Scores (PCS & MCS) and range from 0 to 100. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Functional Impairment | pre-operatively, 6 weeks, 3, 6, 12 and 24 months post operatively
  Questionnaire ODI ( Oswestry Disability Index) - disability questionnaire uses to assess functional impairment of the patient. Regarding lifting, ability to walk, sit, stand sleep, travel graded by score of 0-100 (0 = no disability and 100- maximum disability possible)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kurd, M.D., Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No